CLINICAL TRIAL: NCT00524641
Title: A Patient Follow-up Program to Assess Asthma Control in Patients Using Symbicort® as Maintenance and Relief Therapy in a Single Inhaler (Symbicort® SMART: Budesonide/Formoterol 160/4.5 Mcg, 1 or 2 Inhalations x 2 Times Plus Additional Inhalations as Needed)
Brief Title: Asthma Control-A "Patient Follow up Programme" Maintenance and Reliever Therapy in a Single Inhaler
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Other Study IDs: NIS-RVN-SYM-2007/1; NIS-R84-AST-2007/3
Record Dates: First submitted 2007-08-30; First posted 2007-09-03 (Estimated); Last update posted 2009-07-09 (Estimated); Status verified 2009-07

CONDITIONS: Asthma
Keywords: Asthma; Symbicort; NIS
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To investigate the change in patient's asthma symptom control using ACQ scores after 4 to 6 weeks of Symbicort Turbuhaler (budesonide/ formoterol) in SMART approach.

ELIGIBILITY:
Inclusion Criteria:

* Asthma patients from both sexes, age 18 or older
* Have already been on Symbicort SMART treatment
* Willing to give written informed consents to participate in the program.

Exclusion Criteria:

* Patients who are not willing to give written informed consent
* Patients in emergency care for asthma at ICUs or COPD patients are excluded from the program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital out-patient departments and private clinics in all areas of Vietnam
Sampling Method: Probability Sample
Enrollment: 1254 (Actual)
Dates: Start 2007-07; Primary Completion 2008-03 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dinh Ngoc SY, MD, Study Chair — TB and Lung Disease Hospital, Hanoi; Tran Van Ngoc, MD, PhD, Study Chair — Cho Ray Hospital; Nguyen Hong Duc, Study Chair — Pharm Ngoc Thach Hospital; Do Van Dung, MD, PhD, Study Chair — Ho Chi Minh City Univ of Medicine and Pharmacist
Locations (2):
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City